CLINICAL TRIAL: NCT01879566
Title: Effect of Catheter-based Radiofrequency Ablation Therapy of the Renal Sympathetic-Nerve System for Patient With Sleep Apnea Syndrome and Therapy Resistant Hypertension
Brief Title: Effect of Catheter-based Radiofrequency Ablation Therapy in Patient With Therapy-resistant Hypertension and Sleep Apnea Syndrome
Status: Withdrawn | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: EK2012_0393
Record Dates: First submitted 2013-04-26; First posted 2013-06-18 (Estimated); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Therapy-resistant Hypertension and Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

INTERVENTIONS:
Other: No intervention will be done. The study is observational

SUMMARY:
The aim of this prospective single-center study is to evaluate sympathetic nervous system directly measured by microneurography, 24-hour blood pressure, endothelial function, vascular compliance, quality of life and platelet adhesion in patients with sleep apnea syndrome (defined by a complaint of excessive daytime sleepiness, an Epworth sleepiness score>8[10], and an apnea/hypopnea index (AHI>15/h) before and after catheter-based radiofrequency ablation of renal nerve. If the selected patients are treated with CPAP, this therapy should be stable during the whole study time. Primary and secondary end-point will be measured before and 1, 3, 6 and 12 months after renal sympathetic denervation.

ELIGIBILITY:
Inclusion criteria: We plan to include male or female subjects, age 18-80 with a diagnosis of medium-severe sleep apnea syndrome (defined by symptoms, a complaint of excessive daytime sleepiness, an Epworth sleepiness score >8, and an apnea / hypopnea index >15/h) and a resistant hypertension (systolic blood pressure >140 mmHg or >130 mmHg in patients with type II diabetes or chronic kidney disease, under treatment with three antihypertensive drugs including a diuretic).

If the selected patients are treated with CPAP, this therapy should be stable during the whole study time.

Every patient will be asked for a written informed consent.

Exclusion criteria: - Heart failure (normal ejection fractions on echocardiography and no clinical signs and symptoms of heart failure).

* Long acting nitrates, or PDE-5-Hemmer
* Alcohol or drug abuse,
* Malignancy (unless healed or remission > 5 years)
* Disease with systemic inflammation (e.g. rheumatoid arthritis, M. Crohn)
* Pulmonary Hypertension (PAP>50 mmHg)
* Pregnancy
* Anatomical contraindication to renal denervation
* Know allergy to contrast
* Participation in another study within the last month

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with therapy-resistant arterial hypertension and sleep apnea syndrome
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-05; Primary Completion 2017-04 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Change in sympathetic nervous system activity (burst/min and burst/100 HB) before and after catheter-based radiofrequency ablation | 6 and 12 months
  The primary objective of this study is to evaluate sympathetic nervous system activity in patients with sleep apnea syndrome before and 6 and 12 months after catheter-based radiofrequency ablation therapy of the renal sympathetic-nerve system

SECONDARY OUTCOMES:
Change in 24-hour blood pressure (24 hour, day and night mean) before and after catheter-based renal denervation | 1, 3, 6 12 months
  Change in 24-hour blood pressure (24 hour, day and night mean) before and after catheter-based renal denervation
Change in renal function (creatinin plasma level and GFR CKD-EPI Formula) before and after catheter-based renal denervation | 1, 3, 6, 12
  Change in creatinin plasma level and GFR CKD-EPI Formula before and after catheter-based renal denervation
Change in sleep quality, pulse-oximetry, AHI, quality of life and subjective sleepiness with the Epworth sleepiness score before after catheter-based renal denervation | 1, 3, 6 and 12 months
Change in 24-hour Holter and heart rate variability, echocardiogramm before and after catheter-based renal denervation | 6 and 12 months
Change in vascular function and oxidative stress and inflammation parameters before and after catheter-based renal denervation | 1, 3, 6, and 12 months
  Change in vascular function (endothelial function as flow mediated dilatation, arterial stiffness by pulse wave velocity) and oxidative stress and inflammation parameters before and after catheter-based renal denervation

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Luescher, Professor, MD, Principal Investigator — University Hospital Zurich, Division of Cardiology
Locations (1):
- University Hospital Zurich, Division of Cardiology, Zurich, Canton of Zurich, Switzerland